CLINICAL TRIAL: NCT06276933
Title: A Prospective, Multicenter, Double-blind, Randomized Controlled Study of Camrelizumab Combined With Chemotherapy ± Thalidomide in First-line Treatment of Patients With Advanced NSCLC
Brief Title: A Study of Camrelizumab Combined With Chemotherapy ± Thalidomide in First-line Treatment of Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji University (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Professor, Dongfang Hospital Affiliated to Tongji University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA-NSCLC-II-039
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; Camrelizumab
MeSH Terms: conditions — Lung Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Camrelizumab+Chemotherapy+Thalidomide (Experimental)
  Interventions: Drug: Camrelizumab + chemotherapy+Thalidomide
- Camrelizumab + chemotherapy+placebo (Active Comparator)
  Interventions: Drug: Camrelizumab + chemotherapy+placebo

INTERVENTIONS:
Drug: Camrelizumab + chemotherapy+Thalidomide — Camrelizumab + chemotherapy+Thalidomide Drug: Camrelizumab Camrelizumab 200mg intravenous (IV) on Day 1 of each 21-day cycle，until progression or unacceptable toxicity Other Name: SHR-1210
  Drug: Thalidomide Thalidomide 100mg，po qd； Other Name: Thalidomide
  Drug: Chemotherapy
  Platinum-based chemotherapy:
  Non-small cell lung cancer (non-squamous cell carcinoma): pemetrexed plus carboplatin/cisplatin on Day 1 of each 21-day cycle for 4-6 cycles，pemetrexed every three weeks (Q3W) maintenance for the remainder of the study or until documented PD; Non-small cell lung cancer (squamous cell carcinoma) : paclitaxel/albumin-bound paclitaxel + carboplatin/cisplatin on Day 1 of each 21-day cycle for 4-6 cycles.
  Other Name: Platinum-based chemotherapy
  Arms: Camrelizumab+Chemotherapy+Thalidomide
Drug: Camrelizumab + chemotherapy+placebo — Drug: Camrelizumab Camrelizumab 200mg intravenous (IV) on Day 1 of each 21-day cycle，until progression or unacceptable toxicity Other Name: SHR-1210
  Drug: placebo 100mg placebo 100mg，po qd；
  Drug: Chemotherapy
  Platinum-based chemotherapy:
  Non-small cell lung cancer (non-squamous cell carcinoma): pemetrexed plus carboplatin/cisplatin on Day 1 of each 21-day cycle for 4-6 cycles，pemetrexed every three weeks (Q3W) maintenance for the remainder of the study or until documented PD; Non-small cell lung cancer (squamous cell carcinoma) : paclitaxel/albumin-bound paclitaxel + carboplatin/cisplatin on Day 1 of each 21-day cycle for 4-6 cycles.
  Other Name: Platinum-based chemotherapy
  Arms: Camrelizumab + chemotherapy+placebo

SUMMARY:
To explore and evaluate the safety and efficacy of camrelizumab combined with chemotherapy ± thalidomide in first-line treatment of advanced non-small cell lung cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, both male and female.
2. Histopathology or cytology confirmed advanced Stage IIIB-IV non-small cell lung cancer.
3. No prior systemic treatment to advanced NSCLC . Subjects who have received prior neo-adjuvant, adjuvant chemotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment free interval of at least 12 months from randomization since the last chemotherapy cycle.
4. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
6. Have a life expectancy of at least 3 months.
7. All baseline laboratory requirements will be assessed.
8. Can swallow pills normally.
9. Remission of all acute toxic reactions to previous antitumor therapy to grade 0-1 or to the level specified in the exclusion criteria.
10. Female Subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose, are not breastfeeding, and must be willing to use very efficient barrier methods of contraception for the course of the study through 180 days after the last dose of study treatment. Male subjects whose partners are fertile women should be surgically sterilized or agree to use effective contraception during the trial period and 90 days after the last administration of the study drug, and sperm donation is not allowed during the study period.
11. Subjects has voluntarily agreed to participate by giving written informed consent. Willing and able to follow planned visits, research treatments, laboratory tests and other test procedures.

Exclusion Criteria:

1. Patients with non-small cell lung cancer diagnosed with other histopathological types, including patients with NSCLC containing small cell lung cancer components.
2. Subjects with epidermal growth factor receptor (EGFR)-sensitizing mutation and/or anaplastic lymphoma kinase (ALK) translocation.
3. Patients who have previously received PD-(L)1 or CTLA-4 treatment.
4. Subjects with active CNS metastases are excluded.
5. Subjects with active, known or suspected autoimmune disease. Participants who are in a stable state and do not require systemic immunosuppressive therapy are permitted to enroll.
6. Congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection.
7. Have the following poorly controlled infectious diseases: active viral hepatitis B or C; Have active TB or are currently receiving anti-TB treatment.
8. There is past or present objective evidence of idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, tissue pneumonia (such as bronchitis, vasculitis obliterans), drug-induced pneumonia, active pneumonia on CT examination, or severe impairment of lung function.
9. Subjects with clinically significant cardiovascular and cerebrovascular diseases.
10. Active infection (CTCAE> Grade 2).
11. Diagnosed with immune deficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy not directly related to tumor treatment within 7 days prior to study enrollment; Physiological doses of glucocorticoids are permitted.
12. Other malignancies developed within 5 years prior to admission, excluding adequately treatable cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery.
13. Subjects received major surgery within 4 weeks of the first dose of study treatment or planned during the study period.
14. Subjects had administration of a live, attenuated vaccine within 4 weeks of the first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study.
15. Subjects who are alcohol dependent or have a history of drug or substance abuse within the last 1 year.
16. Subjects with a known neurological or mental disorder, such as epilepsy, dementia, or the presence of a peripheral nervous system disorder.
17. Subjects had or plan to have allogeneic bone marrow transplantation or solid organ transplant.
18. Pregnant or lactating female; The fertile subject is unwilling or unable to take effective contraceptive measures.
19. Known allergy to the investigational drug or excipient.
20. Received any other investigational medicine treatment or participated in another interventional clinical study within 4 weeks prior to signing the ICF.
21. Abnormal coagulation function .Thrombosis or thromboembolic event within 6 months prior to the start of study treatment.
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-02-22 (Estimated); Primary Completion 2025-11-22 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of any grade Reactive Cutaneous Capillary Endothelial Proliferation(RCCEP) | 2 years
  Incidence rate of any grade Reactive Cutaneous Capillary Endothelial Proliferation(RCCEP)

SECONDARY OUTCOMES:
Median time to RCCEP | 2 years
  Median time to RCCEP
Median time to RCCEP of level 3 or above | 2 years
  Median time to RCCEP of level 3 or above
Incidence rate of ≥G3 grade RCCEP | 2 years
  Incidence rate of ≥G3 grade RCCEP
Overall Response Rate (ORR) | 2 years
  Overall Response Rate (ORR)
Progression-Free Survival (PFS) | 2 years
  Progression-Free Survival (PFS)
Overall Survival(OS) | 2 years
  Overall Survival(OS)
Treatment-related Adverse Events (TRAE) | 2 years
  Treatment-related Adverse Events (TRAE)

CONTACTS AND LOCATIONS:
Overall Officials: Anwen Xiong, MD, Study Director — Department of Oncology, Shanghai pulmonary hospital Shanghai, China, 200433

IPD SHARING:
Plan to Share IPD: No